CLINICAL TRIAL: NCT01083901
Title: Acetaminophen and Impaired Musculoskeletal Adaptations to Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 06-0343; R21AG027809 (NIH)
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Sarcopenia; Osteoporosis; Aging
MeSH Terms: conditions — Sarcopenia; Osteoporosis | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resistance training with Acetaminophen (Experimental): Acetaminophen
  Interventions: Behavioral: Resistance training
- Resistance Training with ibuprofen (Experimental): Ibuprofen
  Interventions: Behavioral: Resistance training
- placebo (Placebo Comparator): Placebo
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — high intensity progressive resistance exercise training

SUMMARY:
The purpose of this study is to determine if taking the pain reliever acetaminophen (ACET) interferes with some of the benefits of weight lifting on muscles and bone density in older men.

DETAILED DESCRIPTION:
The commonly used pain relievers acetaminophen and ibuprofen may impair musculoskeletal adaptations to progressive resistance exercise training by inhibiting exercise-induced muscle protein synthesis.

To test the hypothesis that acetaminophen and ibuprofen would diminish training-induced increases in fat-free mass, untrained men (n=26) aged ≥ 50 years participated in 16 weeks of high-intensity progressive resistance exercise training and bone-loading exercises and were randomly assigned to take ACET (1000 mg), ibuprofen (400 mg) or placebo 2 hours before each exercise session.

The primary outcome was the change in total body fat-free mass measured by dual-energy X-ray absorptiometry (DXA) at baseline and week 16. Our primary interest was in the comparison of the acetaminophen and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* average use of acetaminophen and non-steroidal anti-inflammatory drugs (NSAIDs) [including aspirin] less than 3 days per month
* not currently engaged in moderate-to-vigorous weight-lifting exercise
* non-smoker
* willing to participate in a supervised exercise program for 9 months

Exclusion Criteria:

* relative or absolute contraindications to regular use of acetaminophen or NSAIDs including known allergy or intolerance to either drug,history of peptic ulcer or GI bleeding, anemia, asthma with bronchospasm induced by aspirin or other NSAIDS, moderate or severe renal impairment, known hepatobiliary disease
* contraindications to exercise testing and training including congestive heart failure class III or IV, uncontrolled hypertension and unstable cardiovascular disease
* thyroid dysfunction
* orthopedic problems that limit the ability to perform vigorous exercise or increase the likelihood of the use of pain medications
* drugs known to alter bone metabolism
* allergy to lidocaine
* diabetes mellitus requiring pharmacologic therapy

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Jankowski, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from Dec 2006 to Jan 2010. They were recruited from the greater Denver area using advertisements.
Pre-assignment Details: Volunteers who did not meet inclusion criteria were excluded from the study during the initial screening visits prior to randomization to the study arms.
Groups:
- Acetaminophen and Resistance Exercise: Progressive resistance exercise training and bone-loading exercise on up to 6 days per week and administration of acetaminophen, 1000 mg, taken 2 hours before exercise on exercise days for up to 36 weeks.
- Ibuprofen and Resistance Exercise: Progressive resistance exercise training and bone-loading exercise on up to 6 days per week and administration of acetaminophen, 400 mg, taken 2 hours before exercise on exercise days for up to 36 weeks.
- Placebo and Resistance Exercise: Progressive resistance exercise training and bone-loading exercise on up to 6 days per week and placebo pills (matching active study drug) taken 2 hours before exercise on exercise days for up to 36 weeks.
Period: Overall Study
Arm/Group | Acetaminophen and Resistance Exercise | Ibuprofen and Resistance Exercise | Placebo and Resistance Exercise
Started | 13 | 8 | 13
Completed | 12 | 6 | 11
Not Completed | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen and Resistance Exercise | Ibuprofen and Resistance Exercise | Placebo and Resistance Exercise | Total
Number analyzed (Participants) | 13 | 8 | 13 | 34
Age Continuous [Mean (Standard Deviation); unit: years]
  United States | 63 (5) | 58 (6) | 62 (7) | 61 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 13 | 8 | 13 | 34
Height [Mean (Standard Deviation); unit: cm] | 181 (8) | 178 (10) | 176 (7) | 178 (6.4)
Weight [Mean (Standard Deviation); unit: kg] | 94.5 (16.6) | 89.3 (12.5) | 87.9 (18.0) | 90.4 (16.4)
Fat-free mass [Mean (Standard Deviation); unit: kg] — Total body fat-free mass measured by DXA (Hologic Discovery W, version 12.6)
  kg | 65.2 (6.1) | 63.5 (8.2) | 62.7 (9.1) | 63.4 (8.0)
Fat mass [Mean (Standard Deviation); unit: kg] — Total body fat mass measured by DXA (Hologic Discovery W, version 12.6)
  kg | 29.3 (12.6) | 25.8 (5.3) | 25.2 (9.6) | 27.0 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Body Fat-free Mass
Description: change from baseline to 16 weeks in fat-free mass measured by DXA (Hologic Discovery W, version 12.6)
Time Frame: 16 weeks
Population: All participants with baseline and 16 week data were included in the analysis (i.e., intention-to-treat).
Measure: Mean (Standard Error); unit: kg
Arm/Group | Acetaminophen and Resistance Exercise Training | Ibuprofen and Resistance Exercise Training | Placebo and Resistance Exercise Training
Number analyzed (Participants) | 12 | 6 | 11
kg | 1.5 (0.6) | 2.3 (0.9) | 0.7 (0.6)
Statistical Analysis 1: Comparison: Acetaminophen and Resistance Exercise Training vs Ibuprofen and Resistance Exercise Training vs Placebo and Resistance Exercise Training; The null hypothesis was that the changes in total body fat-free mass in response to resistance exercise training would not be different among the groups. The expected difference in fat-free mass between the Acetaminophen and Placebo groups was 1.8 +/- 1.0% with a 3.6 +/1 1.0% increase in fat-free mass in the Placebo group. The study was designed to achieve 96% power at the 0.05 level with 10 men in the acetaminophen and placebo groups; Test type: Superiority or Other; p = 0.38, ANCOVA; Changes from baseline to 16 weeks were regressed on the baseline measurement

2. Secondary Outcome: Change in Total Body Fat Mass
Description: Change from baseline to 16 weeks in total body fat mass.
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: kg
Arm/Group | Acetaminophen and Resistance Exercise Training | Ibuprofen and Resistance Exercise Training | Placebo and Resistance Exercise Training
Number analyzed (Participants) | 12 | 6 | 11
kg | -1.5 (0.6) | -1.4 (0.9) | -0.2 (0.6)
Statistical Analysis 1: Comparison: Acetaminophen and Resistance Exercise Training vs Ibuprofen and Resistance Exercise Training vs Placebo and Resistance Exercise Training; Test type: Superiority or Other; p = 0.23, ANCOVA; The change in fat mass was regressed on the baseline measure

3. Secondary Outcome: Changes in Upper Body Strength.
Description: Strength was measured using the one-repetition maximum method. Upper body strength was a composite of bench press, overhead press, seated row, and lateral pull-down strength.
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: lbs
Arm/Group | Acetaminophen and Resistance Exercise Training | Ibuprofen and Resistance Exercise Training | Placebo and Resistance Exercise Training
Number analyzed (Participants) | 12 | 6 | 11
lbs | 19.5 (5.5) | 35.2 (8.6) | 26.5 (5.8)
Statistical Analysis 1: Comparison: Acetaminophen and Resistance Exercise Training vs Ibuprofen and Resistance Exercise Training vs Placebo and Resistance Exercise Training; Test type: Superiority or Other; p = 0.30, ANCOVA; Change in strength was regressed on baseline measures

4. Secondary Outcome: Change in Lower Body Strength
Description: Strength was measured using the one-repetition maximum method. Lower body strength was a composite of knee flexion, knee extension, and leg press strength.
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: lbs
Arm/Group | Acetaminophen and Resistance Exercise Training | Ibuprofen and Resistance Exercise Training | Placebo and Resistance Exercise Training
Number analyzed (Participants) | 12 | 6 | 11
lbs | 33.1 (9.4) | 40.8 (14.6) | 18.0 (9.8)
Statistical Analysis 1: Comparison: Acetaminophen and Resistance Exercise Training vs Ibuprofen and Resistance Exercise Training vs Placebo and Resistance Exercise Training; Test type: Superiority or Other; p = 0.37, ANCOVA; Changes in strength were regressed on the baseline measure

ADVERSE EVENTS:
Time Frame: Throughout the study.
Arm/Group | Acetaminophen and Resistance Exercise Training | Ibuprofen and Resistance Exercise Traininig | Placebo and Resistance Exercise Training
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/8 | 0/13

LIMITATIONS AND CAVEATS:
This was a preliminary study that was limited by small sample size, exclusion of women, and the duration of intervention which was too brief to measure changes in bone mineral density.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No